CLINICAL TRIAL: NCT01219114
Title: A Descriptive Study of the Efficacy and Safety of CUBICIN (Daptomycin) Under Conditions of Actual Use in the Philippines
Brief Title: Safety and Efficacy Study of CUBICIN (Daptomycin) Under Conditions of Actual Use
Status: Withdrawn | Type: Observational
Why Stopped: Inability to recruit patients within the specified time period. No patients have been enrolled in the study.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-IPH-DUM-2010/1
Record Dates: First submitted 2010-10-10; First posted 2010-10-13 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Complicated Skin and Skin Structure Infections and Bacteremia Including Right-sided Endocarditis
Keywords: Daptomycin; endocarditis; complicated skin and skin structure infection
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to monitor the safety and efficacy of CUBICIN under conditions of actual use in patients who are diagnosed with complicated Skin and Skin Structure infection (cSSI) or Staphylococcus aureus bacteria including right-sided endocarditis and are prescribed CUBICIN by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cSSSI known or suspected to be due to gram-positive bacteria
* Diagnosis of right-sided endocarditis with one or more positive culture for S. aureus within two days prior to initiation of medication
* Prescribed daptomycin by patient's attending physician

Exclusion Criteria:

* Known allergic or serious adverse reaction to daptomycin
* Patients with pneumonia
* Patients with baseline CPK values >1000 U/L or 5x ULN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: several private and government tertiary hospitals
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Adverse events observed during the treatment duration | Ranges from during treatment and up to 14 days after last administration of daptomycin (follow up)
Clinical Response determined by cure rate | Ranges from during treatment and up to 14 days after last administration of daptomycin

CONTACTS AND LOCATIONS:
Overall Officials: Milagros Tan, MD, Study Director — AstraZeneca Philippines; Emmanuel Arca, MD, Study Chair — AstraZeneca Philippines
Locations (5):
- Philippines (5):
  - Research Site, Lipa City, Batangas
  - Research Site, Davao City, Davao Region
  - Research Site, Iloilo City, Iloilo
  - Research Site, Pasig, National Capital Region
  - Research Site, Quezon City, National Capital Region